CLINICAL TRIAL: NCT03414034
Title: A Phase 2 Study of PCM-075 (Onvansertib) in Combination With Abiraterone and Prednisone in Adult Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Onvansertib in Combination With Abiraterone and Prednisone in Adult Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TROV-053; U1111-1208-1579 (Registry Identifier: WHO)
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: PLK1; PLK Inhibitor; Onvansertib
MeSH Terms: interventions — onvansertib; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: onvansertib + abiraterone and prednisone (Experimental): On Day 1 of each cycle, onvansertib will be administered orally (PO) once daily (QD) at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 21-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants will also receive abiraterone and prednisone. This arm was discontinued.
  Interventions: Drug: Onvansertib; Drug: Abiraterone; Drug: Prednisone
- Arm B: onvansertib + abiraterone and prednisone (Experimental): On Day 1 of each cycle, onvansertib will be administered orally (PO) once daily (QD) at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants will also receive abiraterone and prednisone.
  Interventions: Drug: Onvansertib; Drug: Abiraterone; Drug: Prednisone
- Arm C: onvansertib + abiraterone and prednisone (Experimental): On Day 1 of each cycle, onvansertib will be administered orally (PO) once daily (QD) at a dose of 12 mg/m^2 for 14 days (Day 1 through Day 14) out of a 21-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants will also receive abiraterone and prednisone.
  Interventions: Drug: Onvansertib; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Onvansertib — Onvansertib orally
  Other Names: PCM-075
Drug: Abiraterone — Abiraterone orally
Drug: Prednisone — Prednisone orally

SUMMARY:
The purpose of the phase 2 study is to determine whether Onvansertib is safe and tolerable in adult participants with Metastatic Castration-Resistant Prostate Cancer who have disease progression while receiving abiraterone acetate (abiraterone) and prednisone therapy, and to observe the effects of Onvansertib in combination with abiraterone and prednisone on disease control.

ELIGIBILITY:
Inclusion Criteria:

1. Males ≥ 18 years of age on the day of consenting to the study.
2. Ability to swallow the study drug as a whole tablet.
3. Histologically confirmed prostate adenocarcinoma without significant small- cell/neuroendocrine or other variant histologies, with rising PSA and/or radiographic progression in the setting of castration-level testosterone (< 50 ng/dL) indicating mCRPC. Participants must have either undergone surgical castration or continue on GnRH agonist/antagonist on the appropriate schedule throughout the study period.
4. Asymptomatic or minimally symptomatic disease.
5. Metastatic disease by bone scan or other nodal or visceral lesions on CT or MRI at any time (past or present).
6. Participant currently receiving abiraterone and prednisone for CRPC.
7. Participant has been on abiraterone for castration-sensitive prostate cancer (CSPC) or castration-resistant prostate cancer (CRPC). Participants who have received abiraterone for CSPC must have had a response to hormonal therapy, as defined by any decline in PSA, radiographic response and/or clinical benefit after starting hormonal therapy.

   Participants who have received abiraterone for CRPC must have responded to abiraterone, defined by any decline in PSA, radiographic response, and/or clinical benefit after starting abiraterone.
8. Two rising PSA values separated by at least 1 week, one showing a rise of at least 0.3 ng/mL and one confirmatory value not showing a decline, while on abiraterone therapy.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
10. Participant has adequate bone marrow and organ function as shown by:

    * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L
    * Platelets ≥ 100 x 10^9/L
    * Hemoglobin (Hgb) ≥ 9.0 g/dL
    * Serum creatinine ≤ 2 x the upper limit of normal (ULN)
    * Total serum bilirubin ≤ 1.5 x ULN (in participants with known Gilbert Syndrome, a total bilirubin ≤ 3.0 x ULN, with direct bilirubin ≤ 1.5 x ULN)
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN (or ≤ 5.0 x ULN if hepatic metastases are present)

Exclusion Criteria:

1. Major surgery within 28 days prior to starting study drug or has not recovered from major side effects of the surgery.
2. Rapidly progressive symptoms of mCRPC.
3. Acute neurological dysfunction as a result of bone metastasis.
4. Previously treated with enzalutamide or experimental therapies directed against androgen receptor (ie, apalutamide).
5. Use of any chemotherapy, investigational agents, immunotherapy, or hormonal therapy other than GnRH agonists within 28 days of the start of treatment on protocol.

   Use of bone targeted agents including bisphosphonates and RANK ligand inhibitors is allowed if on stable dose; Xgeva or Zometa cannot be started within 28 days of initiating study therapy.
6. Systemic corticosteroids except as part of on label treatment prostate cancer regimens. Note: Topical applications (eg, rash), inhaled sprays (eg, obstructive airways diseases), eye drops or local injections (eg, intra-articular) are allowed.
7. Treatment with any of the drugs listed in Section 8.4.5 at the time of study treatment initiation.
8. Has received wide field radiotherapy (including therapeutic radioisotopes such as radium 223) ≤ 28 days or limited field radiation for palliation ≤ 14 days prior to starting study drug or has not recovered from side effects of such therapy.
9. New York Heart Association (NYHA) Class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition, or hypertensive or metabolic condition.
10. Myocardial infarction in the previous 12 weeks (from the start of treatment)
11. QT interval with Fridericia's correction [QTcF] >470 milliseconds. The QTcF should be calculated as the arithmetic mean of the QTcF on triplicate ECGs. In the case of potentially correctible causes of QT prolongation (e.g., medications, hypokalemia), the triplicate ECG may be repeated once during screening and that result may be used to determine eligibility.
12. Planned concomitant use of medications known to prolong the QT/QTc interval
13. Presence of risk factors for torsade de pointes, including family history of Long QT Syndrome or uncorrected hypokalemia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hagege A, Ambrosetti D, Boyer J, Bozec A, Doyen J, Chamorey E, He X, Bourget I, Rousset J, Saada E, Rastoin O, Parola J, Luciano F, Cao Y, Pages G, Dufies M. The Polo-like kinase 1 inhibitor onvansertib represents a relevant treatment for head and neck squamous cell carcinoma resistant to cisplatin and radiotherapy. Theranostics. 2021 Sep 21;11(19):9571-9586. doi: 10.7150/thno.61711. eCollection 2021. PMID 34646387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 participants with Metastatic Castration-Resistant Prostate Cancer (mCRPC) were enrolled at 3 investigative sites in the United States between August 2018 and October 2023. Arm A was discontinued with Protocol Version 1.6 (08 Nov 2019). Any participants enrolled and were continuing treatment in Arm A had the opportunity to transition to Arm B (with a re-consent) at the start of their next cycle and at the discretion of the Investigator.
Groups:
- Arm A: Onvansertib + Abiraterone and Prednisone: On Day 1 of each cycle, onvansertib was administered orally (PO), once daily (QD) at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 21-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone. This arm was discontinued.
- Arm B: Onvansertib + Abiraterone and Prednisone: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle. Following dose limiting toxicity (DLT), the final recommended dose was reduced to 18 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle as pre-specified in the protocol. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone.
- Arm C: Onvansertib + Abiraterone and Prednisone: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 12 mg/m^2 for 14 days (Day 1 through Day 14) out of a 21-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone.
Period: Overall Study
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Started | 24 | 20 | 28
Transferred to Arm B | 2 | 0 (Not applicable to this arm.) | 0 (Not applicable to this arm.)
Completed | 0 | 0 | 0
Not Completed | 24 | 20 | 28
Not completed — Adverse Event | 6 | 1 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Non-compliance With Study Drug | 0 | 0 | 1
Not completed — Physician Decision | 1 | 3 | 2
Not completed — Withdrawal of Informed Consent | 2 | 1 | 4
Not completed — Progressive Disease | 15 | 15 | 17
Not completed — Miscellaneous | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population: comprises all participants who received any dose of onvansertib.
Groups:
- Arm A: Onvansertib + Abiraterone and Prednisone: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 21-day cycle. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone. This arm was discontinued.
- Arm B: Onvansertib + Abiraterone and Prednisone: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle. Following DLT, the final recommended dose was reduced to 18 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle as pre-specified in the protocol. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone.
- Total: Total of all reporting groups
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone | Total
Number analyzed (Participants) | 24 | 20 | 28 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.44) | 71.3 (8.39) | 69.4 (9.12) | 70.4 (8.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 24 | 20 | 28 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 16 | 25 | 61
  Unknown or Not Reported | 4 | 3 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Black or African American | 0 | 3 | 2 | 5
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  White | 24 | 17 | 23 | 64
  Other | 0 | 0 | 1 | 1
  Unknown | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Disease Control at or Before 12 Weeks
Description: Disease control was defined as lack of prostate-specific antigen (PSA) progression per Prostate Cancer Working Group 3 (PCWG3) criteria: not having an increase in PSA from Baseline or nadir ≥ 25% and ≥ 2 ng/mL during the first 12 weeks of PSA assessments. Participants that do not have 12 weeks of PSA assessments were considered not to have demonstrated PSA progression control in this analysis. If a participant achieved disease control prior to Week 12, but relapsed at, or before Week 12, disease control was still considered achieved. The 90% confidence intervals were calculated using Wilson Confidence Interval.
Time Frame: Baseline up to Week 12
Population: Efficacy Population: comprises all participants who received at least 1 dose of onvansertib at the final recommended dose according to their arm assignments. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm A to B: Onvansertib + Abiraterone and Prednisone: Arm A: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 21-day cycle.
  Following discontinuation of Arm A, participants transferred to Arm B: On Day 1 of each cycle, onvansertib was administered PO, QD at a dose of 24 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle. Following DLT, the final recommended dose was reduced to 18 mg/m^2 for 5 days (Day 1 through Day 5) out of a 14-day cycle as pre-specified in the protocol.
  Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone.
- Total: Inclusive of participants enrolled in Arms A, A to B, B, and C.
  On Day 1 of each cycle, onvansertib was administered PO, QD. Beginning on Day 1 and continuing uninterrupted throughout each cycle, participants also received abiraterone and prednisone.
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone | Total
Number analyzed (Participants) | 22 | 2 | 20 | 28 | 72
percentage of participants | 13.6 [5.6 to 29.7] | 50.0 [12.1 to 87.9] | 35.0 [20.2 to 53.3] | 35.7 [22.7 to 51.3] | 29.2 [21.2 to 38.6]

2. Secondary Outcome: Mean Percentage Change From Baseline in PSA at 12 Weeks
Description: PSA level was measured via blood sample. Mean and standard deviation change is reported.
Time Frame: Baseline and Week 12
Population: 100% Per-protocol (PP) Population: consists of participants who have been administered 100% of the originally assigned study drugs in at least one full cycle, and without major protocol deviations. If a participant did not have a Week 12 (+/- 3 days) PSA measure, then they are not included in this analysis. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Mean (Standard Deviation); unit: percentage of PSA
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 8 | 2 | 12 | 21
percentage of PSA | 84.330 (52.545) | 67.064 (50.350) | 42.661 (60.818) | 77.675 (94.611)

3. Secondary Outcome: Mean Absolute Change From Baseline in PSA at 12 Weeks
Description: PSA level was measured via blood sample. Mean and standard deviation change is reported.
Time Frame: Baseline and Week 12
Population: 100% PP Population: consists of participants who have been administered 100% of the originally assigned study drugs in at least one full cycle, and without major protocol deviations. If a participant did not have a Week 12 (+/- 3 days) PSA measure, then they are not included in this analysis. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 8 | 2 | 12 | 21
ng/mL | 10.904 (10.141) | 3.095 (2.199) | 14.971 (45.023) | 7.295 (13.076)

4. Secondary Outcome: Median Percentage Change From Baseline in PSA at 12 Weeks
Description: PSA level was measured via blood sample. Median, minimum and maximum change is reported.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of PSA
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 8 | 2 | 12 | 21
percentage of PSA | 94.814 [8.443 to 155.720] | 67.064 [31.461 to 102.667] | 25.828 [-65.823 to 137.069] | 54.630 [-31.414 to 401.348]

5. Secondary Outcome: Median Absolute Change From Baseline in PSA at 12 Weeks
Description: PSA level was measured via blood sample. Median, minimum and maximum change is reported.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 8 | 2 | 12 | 21
ng/mL | 9.110 [0.19 to 26.00] | 3.095 [1.54 to 4.65] | 1.345 [-20.80 to 155.00] | 2.300 [-5.73 to 47.64]

6. Secondary Outcome: Time to PSA Progression or Death
Description: Time to PSA progression in weeks is defined as time from Cycle 1 Day 1 (initiation of treatment) until initiation of any PSA progression per PCWG3 criteria: an increase in PSA from Baseline or nadir ≥ 25% and ≥ 2 ng/mL. If a participant discontinued from the study without confirmed PSA progression or death, then they were censored at the last PSA laboratory date. Kaplan-Meier method was used.
Time Frame: Up to approximately 100 weeks
Population: 100% PP Population: consists of participants who have been administered 100% of the originally assigned study drugs in at least one full cycle, and without major protocol deviations. Only participants with available data are included in the analysis. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 15 | 2 | 18 | 25
weeks | 5.1 [3.0 to 9.0] | 10.5 [3.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 10.9 [4.0 to 18.0] | 9.0 [8.0 to 18.0]

7. Secondary Outcome: Time to Radiographic Progression or Death
Description: Time to radiographic progression in weeks is defined as time from Cycle 1 Day 1 (initiation of treatment) until initiation of any radiographic progression per PCWG3 criteria. If a participant discontinued from the study without confirmed radiographic progression or death, then they were censored at the last valid assessment date.
Time Frame: Up to approximately 110 weeks
Population: 100% PP Population: consists of participants who have been administered 100% of the originally assigned study drugs in at least one full cycle, and without major protocol deviations. Only participants with target or non-target lesions at Baseline are included in the analysis. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 15 | 2 | 18 | 25
weeks | 12.0 [8.6 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | NA [NA to NA] — Median and confidence intervals were not calculable due to insufficient events (0). | 17.4 [3.9 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 57.0 [19.1 to 96.1]

8. Secondary Outcome: Percentage of Participants Achieving Radiographic Responses at or Before 12 Weeks
Description: Radiographic response is defined as the best overall response between Cycle 1 Day 1 and 12 weeks post-baseline being stable disease (SD) or better (partial response [PR] or complete response [CR]) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1):
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD).
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: Baseline up to Week 12
Population: 100% PP Population: consists of participants who have been administered 100% of the originally assigned study drugs in at least one full cycle, and without major protocol deviations. Only participants with target or non-target lesions at Baseline and at least 1 post-baseline assessment are included. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 7 | 0 | 8 | 10
percentage of participants | 28.6 [10.0 to 59.1] |  | 62.5 [34.8 to 83.9] | 80.0 [54.1 to 93.1]

9. Secondary Outcome: Percentage of Participants Who Are Adherent to Study Treatment (PP Analysis) Achieving Disease Control at or Before 12 Weeks
Description: Disease control was defined as lack of PSA progression per PCWG3 criteria: not having an increase in PSA from Baseline or nadir ≥ 25% and ≥ 2 ng/mL during the first 12 weeks of PSA assessments. Participants that do not have 12 weeks of PSA assessments were considered not to have demonstrated PSA progression control in this analysis. If a participant achieved disease control prior to Week 12, but relapsed at, or before Week 12, disease control was still considered achieved. The 90% confidence intervals were calculated using Wilson Confidence Interval.
Time Frame: Baseline up to Week 12
Population: as for outcome 6
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 15 | 2 | 18 | 25
percentage of participants | 13.3 [4.5 to 33.4] | 50.0 [12.1 to 87.9] | 38.9 [22.7 to 58.0] | 36.0 [22.3 to 52.4]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse events (AEs) are defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. TEAEs are defined as AEs with a start date after Cycle 1 Day 1. AE severity was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 on a scale from Grade 1 (mild) to Grade 5 (death related to AE).
Time Frame: Up to approximately 27 months
Population: Safety Population: comprises all participants who received any dose of onvansertib. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 22 | 2 | 20 | 28
Participants
  Any TEAEs | 22 | 2 | 20 | 27
  Any TEAEs with CTCAE Grade ≥3 | 12 | 0 | 11 | 13

11. Secondary Outcome: Number of Participants With DLTs
Description: DLTs are defined as a CTCAE Grade 4 hematologic AE or CTCAE Grade ≥ 3 non-hematologic AE that is considered related to the study drug.
Time Frame: Arms A and B: up to one 21-day cycle; Arm C: up to two 14-day cycles
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
Number analyzed (Participants) | 22 | 2 | 20 | 28
Participants | 4 | 0 | 4 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: Safety Population: comprises all participants who received any dose of onvansertib. Arm A participants who transferred to Arm B and those who did not transfer are summarized separately.
Arm/Group | Arm A: Onvansertib + Abiraterone and Prednisone | Arm A to B: Onvansertib + Abiraterone and Prednisone | Arm B: Onvansertib + Abiraterone and Prednisone | Arm C: Onvansertib + Abiraterone and Prednisone
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/2 | 0/20 | 2/28
Serious Adverse Events (participants affected / at risk) | 5/22 | 0/2 | 5/20 | 6/28
Other Adverse Events (participants affected / at risk) | 21/22 | 2/2 | 20/20 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Onvansertib + Abiraterone and Prednisone (N=22) | Arm A to B: Onvansertib + Abiraterone and Prednisone (N=2) | Arm B: Onvansertib + Abiraterone and Prednisone (N=20) | Arm C: Onvansertib + Abiraterone and Prednisone (N=28)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 3
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Onvansertib + Abiraterone and Prednisone (N=22) | Arm A to B: Onvansertib + Abiraterone and Prednisone (N=2) | Arm B: Onvansertib + Abiraterone and Prednisone (N=20) | Arm C: Onvansertib + Abiraterone and Prednisone (N=28)
Anaemia (Blood and lymphatic system disorders) | 8 | 1 | 8 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 0 | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 8 | 0 | 8 | 5
Leukopenia (Blood and lymphatic system disorders) | 5 | 0 | 4 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 6
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 11 | 1 | 6 | 10
Oedema peripheral (General disorders) | 2 | 0 | 2 | 2
Chills (General disorders) | 1 | 0 | 2 | 1
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 2 | 0
Malaise (General disorders) | 1 | 0 | 0 | 1
Hernia (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 1 | 9 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 6 | 5
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 3 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 5
Constipation (Gastrointestinal disorders) | 3 | 0 | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0 | 2 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 0 | 1 | 0
Eyelid infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 5
Blood creatinine increased (Investigations) | 2 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Bronchial wall thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 5 | 6
Hot flush (Vascular disorders) | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 5 | 1
Headache (Nervous system disorders) | 1 | 0 | 3 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vasculitic rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-11-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT03414034/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT03414034/SAP_001.pdf